CLINICAL TRIAL: NCT00120159
Title: GPRN Neonatal Surgical Database: Necrotizing Enterocolitis (NEC) Protocol
Brief Title: Necrotizing Enterocolitis (NEC) Surgical Database
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Glaser Pediatric Research Network (Network); Elizabeth Glaser Pediatric AIDS Foundation (Other); Yale University (Other)
Other Study IDs: X03-12-080
Record Dates: First submitted 2005-06-30; First posted 2005-07-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2006-01

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The general objectives of this protocol are to develop a multi-center prospective data collection process to identify risk factors for progression of Necrotizing Enterocolitis (NEC). These data will be used as a basis for identifying management strategies appropriate for further evaluation (randomized controlled trials), to develop evidence-based standards of care, and as a tool to facilitate quality-assessment at individual centers through comparison of outcomes with the entire database.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet at least one criterion from each of the following three categories:

Historical Factors:

* Feeding intolerance defined as vomiting of 2 or more feedings within 24 hours or any vomitus containing bile, or the presence of gastric residuals of volume greater than 6cc/kg or any aspirate containing bile
* Apneic/bradycardic episodes
* Oxygen desaturation episode not otherwise explained
* Guaiac positive or grossly bloody stools

Physical Examination Findings:

* Abdominal distention recorded by practitioner
* Capillary refill time greater than 2 seconds
* Abdominal wall discoloration
* Abdominal tenderness

Radiographic Findings:

* Pneumatosis intestinalis
* Portal venous gas
* Ileus
* Dilated bowel
* Pneumoperitoneum
* Air/fluid levels
* Thickened bowel walls
* Ascites or peritoneal fluid
* Free intraperitoneal air

Exclusion Criteria:

Patients will be excluded for any of the following:

* Major gastrointestinal anomaly
* Prior abdominal operation
* Family does not consent to participate (A list of patients for whom consent was refused will be maintained in order to avoid contacting these families repeatedly. All families who refuse consent will be queried as to the reason for refusal).

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Tom Jaskic, MPH, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States